CLINICAL TRIAL: NCT04815928
Title: Registry of Patients That Have Undergone an Invasive Coronary Angiography and/or Percutaneous Coronary Intervention
Brief Title: Registry of Patients That Have Undergone ICA or PCI
Acronym: ICA-PI
Status: Recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Paul Knaapen, Principal Investigator, Amsterdam UMC, location VUmc
Other Study IDs: ICA-PI
Record Dates: First submitted 2021-03-18; First posted 2021-03-25 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Coronary Artery Disease
Keywords: Quantiative Flow Ratio; QFR; Fractional Flow Reserve; FFR; Instantaneous wave-free ratio; iFR; Invasive Coronary Angiography; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In Invasive Coronary Angiography there are multiple invasively obtained measurements to determine the funcitonal significance of Cornary Artery Disease. In this Registry, patients who have undergone Invasive Coronary Angiography or Percutaneous Coronary Intervention are included to investigate diagnostic and prognostic implications of the invasive measurements.

ELIGIBILITY:
Inclusion Criteria:

* 18 years
* Has undergone or will undergo a clinically indicated invasive coronary angiography.
* Has undergone or will undergo a clinically indicated percutaneous coronary intervention.

Exclusion Criteria:

* Not willing / unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that have undergone an invasive coronary angiography and or/percutaneous coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2035-07-01 (Estimated); Study Completion 2035-07-01 (Estimated)

PRIMARY OUTCOMES:
Fractional Flow Reserve (FFR) | Upon inclusion at index procedure
  Invasively obtained FFR
Instantaneous wave-free ratio (iFR) | Upon inclusion at index procedure
  Invasively obtained iFR
Quantitative Flow Ratio (QFR) | Upon inclusion at index procedure
  Invasively obtained QFR
Stenosis percentage | Upon inclusion at index procedure
  Invasively obtained stenosis percentage

SECONDARY OUTCOMES:
Major adverse cardiac events, cardiac death or repeat revascularization | 5 years
  The secondary endpoint is to assess the prognostic value of the obtained parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam Univeristy Medical centers, location VUmc, Amsterdam, Netherlands